CLINICAL TRIAL: NCT01019512
Title: A Pilot, Randomized, Single-Blind Study to Assess the Efficacy of the FlexitouchÂ® Lymphedema System in Reducing Lymphedema in Patients Treated for Breast Cancer
Brief Title: Flexitouch Lymphedema System in Treating Stage II Lymphedema in Patients With Breast Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Alavi, Abass, Abramson Cancer Center of The University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: UPCC 02109; NCI-2009-01415
Record Dates: First submitted 2009-11-23; First posted 2009-11-24 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2015-03

CONDITIONS: Breast Cancer; Lymphedema
MeSH Terms: conditions — Breast Neoplasms; Lymphedema

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm I (Active Comparator): Patients undergo complex decongestive therapy comprising daily compression garment (sleeve and glove) use, daily manual lymphatic drainage (self-administerd), and nighttime bandaging with low stretch Comprilan bandages.
  Interventions: Other: questionnaire administration; Other: lymphedema management
- Arm II (Experimental): Patients undergo daily compression with garments (sleeve and glove), nighttime bandaging with low stretch Comprilan bandages, and daily Flexitouch treatment over 1 hour every evening.
  Interventions: Other: questionnaire administration; Other: lymphedema management
- Arm III (Experimental): Patients undergo daily compression with garments (sleeve and glove) and daily Flexitouch treatment over 1 hour every evening.
  Interventions: Other: questionnaire administration; Other: lymphedema management

INTERVENTIONS:
Other: questionnaire administration — Ancillary studies
Other: lymphedema management

SUMMARY:
RATIONALE: The Flexitouch lymphedema system may lessen lymphedema caused by treatment for breast cancer. It is not yet known whether the Flexitouch lymphedema system is more effective than complex decongestive therapy in treating lymphedema. PURPOSE: This randomized clinical trial is studying the Flexitouch lymphedema system in treating stage II lymphedema in patients with breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES: I. To quantitatively assess, by circumferential measurements and CT imaging techniques, the ability of the Flexitouch Lymphedema System to maintain reductions in limb volume after completion of the reductive phase of complex decongestive therapy in a population of patients with upper limb lymphedema secondary to the effects of breast cancer treatment. SECONDARY OBJECTIVES: I. To determine the drainage territory of the lymphatics of the affected arm and chest using CT and to determine whether these patterns are changed by treatment with the Flexitouch Lymphedema System/daytime garments versus Flexitouch Lymphedema System/daytime garments/nighttime bandaging versus standard self-care. OUTLINE: Patients are randomized to 1 of 3 treatment arms. Arm I: Patients undergo complex decongestive therapy comprising daily compression garment (sleeve and glove) use, daily manual lymphatic drainage (self-administered), and nighttime bandaging with low stretch Comprilan bandages. Arm II: Patients undergo daily compression with garments (sleeve and glove), nighttime bandaging with low stretch Comprilan bandages, and daily Flexitouch treatment over 1 hour every evening. Arm III: Patients undergo daily compression with garments (sleeve and glove) and daily Flexitouch treatment over 1 hour every evening. In all arms, treatment continues for 3 months.

ELIGIBILITY:
Inclusion

* Subjects must have a known, clinical diagnosis of stage II lymphedema as verified by a physician specializing in this disorder
* Subjects must have had a unilateral mastectomy, lymph node (LN) dissection and/or radiation therapy for the treatment of primary breast cancer
* Subjects must have completed their course of adjuvant chemotherapy
* Clinical assessment of lymphedema demonstrating at least 10% difference between the volumes of the affected and opposite limbs at the time of enrollment
* Subjects must be completing phase I of their CDT for their initial onset of lymphedema or for an acute flare of lymphedema
* Subjects must be capable of giving informed consent Exclusion
* History of prior trauma and/or surgery in the affected limb other than that for treatment of breast cancer
* Patients with recurrent breast cancer
* History of bilateral breast cancer
* Subjects currently receiving other therapies for lymphedema
* Subjects with renal, liver, and/or heart dysfunction
* Open wounds or web syndrome
* Active/acute infection (cellulitis)
* Acute DVT/Thrombophlebitis
* Decompensated or untreated congestive heart failure
* Pulmonary embolism - Pregnancy as confirmed by urine test; all patients of child bearing potential will be required to have a urine pregnancy test
* Subjects cannot be homeless persons
* Concomitant chemotherapy and radiation treatment during this study is not permitted

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2009-07; Primary Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Upper extremity volume measured by circumferential measurements and by CT imaging | At baseline, monthly for 3 months (circumferential measurements only), and end of study
Signs and symptoms of acute infection

SECONDARY OUTCOMES:
Weight | At baseline and then monthly for 3 months
BMI | At baseline and then monthly for 3 months
Upper body function, based on the Disability of Arm, Shoulder, and Hand Scale (DASH) | At baseline and then monthly for 3 months
Functional assessment, based on the Functional Assessment of Cancer Therapy Breast + 4 (FACT+4) | At baseline and then monthly for 3 months
Quality of life, based on the Functional Assessment of Cancer Therapy Breast (FACT-B) | At baseline and then monthly for 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Abass Alavi, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of The University of Pennsylvania, Philadelphia, Pennsylvania, United States